CLINICAL TRIAL: NCT02809313
Title: Clinical and Microbiological Effects of Lactobacillus Rhamnosus in Treatment of Gingivitis: a Randomized Placebo-controlled Trials With 3-month Follow-up
Brief Title: Clinical and Microbiological Effects of Lactobacillus Rhamnosus in Treatment of Gingivitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jorge Gamonal (Other)
Responsible Party: Sponsor-Investigator, Jorge Gamonal, Professor, University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1130570
Record Dates: First submitted 2016-06-13; First posted 2016-06-22 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-06

CONDITIONS: Gingivitis
Keywords: gingivitis; probiotic; non- surgical treatment
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Gingivitis with Probiotic (Experimental): Gingivitis group of patient treated with conventional therapy (scaling, coronary polish and oral hygiene instruction) and adjunct probiotic containing one sachet Lactobacillus rhamnosus per day during 3 month
  Interventions: Dietary Supplement: Treatment Gingivitis with Probiotic
- Treatment Gingivitis conventional (Placebo Comparator): Gingivitis group of patient treated with conventional therapy (scaling, coronary polish and oral hygiene instruction) and adjunct placebo containing one sachet placebo (talc power) per day during 3 month
  Interventions: Other: Treatment Gingivitis conventional

INTERVENTIONS:
Dietary Supplement: Treatment Gingivitis with Probiotic — gingivitis treatment (scaling and coronary polish) and one sachet containing Lactobacillus rhamnosus SP1 per day during 3 months
  Arms: Treatment Gingivitis with Probiotic
Other: Treatment Gingivitis conventional — gingivitis treatment (scaling and coronary polish) and one sachet containing Placebo (talc powder) per day during 3 months
  Arms: Treatment Gingivitis conventional

SUMMARY:
The aim of this randomized placebo- controlled clinical trial is to evaluate the effects of Lactobacillus rhamnosus SP1- containing probiotic sachet as an adjunct to scaling and root planning (SRP). Material and methods: Thirty six gingivitis patients will be recruited and monitored clinically and microbiologically at baseline and 3-6 months after therapy. All patients will receive scaling and periodontal treatment and randomly will be assigned over an experimental (SRP + probiotic, n=18) or control (SRP + placebo, n=18) group. The sachet will be used once per day during 3 months.

DETAILED DESCRIPTION:
Gingivitis is the most prevalent worldwide periodontal disease, is characterized by inflammation of the tissues surrounding the tooth without causing periodontal attachment loss. Preventive and / or therapeutic measures to facilitate or improve their control are therefore very important, much more if you consider that gingivitis and periodontitis are considered part of an ongoing inflammatory process. Treatment of gingivitis, like that of all periodontal diseases has been based on the implementation of control measures personal and professional plaque. Notwithstanding the foregoing, it has been reported that although mechanical therapy achieved significantly decrease the periodontopathogens, this may be only temporary since bacteria can recolonize the treated niches in the oral cavity. In this context, it has emerged as a new treatment strategy complementary use of probiotics such as Lactobacillus rhamnosus, which possess anti-bacterial and anti-inflammatory properties. Generally speaking, probiotics would promote health by competitive exclusion of some or positive pathogenic bacteria. Objective: To evaluate the effect of the administration of Lactobacillus rhamnosus as an adjunct to conventional periodontal therapy in adolescent and young adult patients with gingivitis. Methodology: A randomized double-blind clinical trial to evaluate the effect of sachet probiotic Lactobacillus rhamnosus as an adjunct to conventional periodontal treatment of patients with gingivitis will be performed. Expected Results: Statistically significant decrease in levels of periodontopathogens (P. gingivalis, A. actinomycetemcomitans, T. forsythia and A. viscosus) in the experimental group compared with the control. Association between clinical and microbiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gingivitis
* Gingival index > 1.5 (> 10 % of the sites examined)
* Index increased bleeding on probing 10% of the sites surveyed
* Probing Depth < 3 mm
* Systemically healthy (except for the presence of gingivitis)
* Patients who have not received periodontal treatment and before no intake of medicines such as antibiotics and / or anti-inflammatory in the last 3 months prior to the start of the study

Exclusion Criteria:

* Patients who develop systemic disease during the study.
* Patients who have to ingest antibiotics and / or antiinflammatories during the study.
* If you are a woman becomes pregnant during the study.

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Differences between groups for bleeding on probing changes | baseline, 3 month, 6 month

SECONDARY OUTCOMES:
Differences between groups for gingival index | baseline, 3 month, 6 month
Differences between groups for detection of periodontal pathogens | baseline, 3 month, 6 month
  P. gingivalis, A. actinomicetemcomitans, T. forsythia and A. viscosus
Differences between groups for levels of periodontal pathogens changes | baseline, 3 month, 6 month
  P. gingivalis, A. actinomicetemcomitans, T. forsythia and A. viscosus

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gamonal Aravena, Proffesor, Principal Investigator — Faculty of Dentistry of University of Chile
Locations (1):
- Faculty of Dentistry of University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No